CLINICAL TRIAL: NCT02173223
Title: A Prospective Study to Assess the Hypotensive Efficacy of Rho-Kinase Inhibitor AR-12286 Ophthalmic Solution 0.5% and 0.7% in Patients With Uncontrolled Advanced Glaucoma With Prior Failed Trabeculectomy or Tube Shunt
Brief Title: A Study to Assess the Effect of Rho-Kinase Inhibitor AR-12286 Ophthalmic Solution 0.5% and 0.7% in Patients With Uncontrolled Advanced Glaucoma With Prior Failed Trabeculectomy or Tube Shunt
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Glaucoma Research Institute (Other)
Responsible Party: Principal Investigator, Jessica Jasien, Co-Investigator, New York Glaucoma Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14.14
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Advanced Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 0.7% Rho-Kinase Inhibitor (Experimental): AR-12286 is a novel Rho-kinase inhibitor developed by Aerie Pharmaceuticals, Inc., Bridgewater, NJ. It is a potent Rho-kinase inhibitor with single-digit nanomolar inhibitory activity against Rho-kinase in enzymatic inhibition assays (deLong MA, et al. IOVS 2009; 50: ARVO E-abstract 4058). Mechanism-of action studies in monkeys demonstrate that AR-12286 lowers IOP primarily by increasing aqueous humor outflow through the trabecular meshwork (Wang RF, et al. IOVS 2009; 50:ARVO E-abstract 1465). Rho-kinase AR-12286 is well tolerated and produces clinically and statistically significant ocular hypotensive efficacy in patients with ocular hypertension and glaucoma. It is well tolerated by most of patients and the only side effect was ocular hyperemia in a minority of subjects (Williams, Novack, Van Haarlem, & Kopczynski, 2011). It is currently in phase II testing.
  Interventions: Drug: Rho-Kinase Inhibitor
- 0.5% Rho-Kinase Inhibitor (Experimental): AR-12286 is a novel Rho-kinase inhibitor developed by Aerie Pharmaceuticals, Inc., Bridgewater, NJ. It is a potent Rho-kinase inhibitor with single-digit nanomolar inhibitory activity against Rho-kinase in enzymatic inhibition assays (deLong MA, et al. IOVS 2009; 50: ARVO E-abstract 4058). Mechanism-of action studies in monkeys demonstrate that AR-12286 lowers IOP primarily by increasing aqueous humor outflow through the trabecular meshwork (Wang RF, et al. IOVS 2009; 50:ARVO E-abstract 1465). Rho-kinase AR-12286 is well tolerated and produces clinically and statistically significant ocular hypotensive efficacy in patients with ocular hypertension and glaucoma. It is well tolerated by most of patients and the only side effect was ocular hyperemia in a minority of subjects (Williams, Novack, Van Haarlem, & Kopczynski, 2011). It is currently in phase II testing.
  Interventions: Drug: Rho-Kinase Inhibitor

INTERVENTIONS:
Drug: Rho-Kinase Inhibitor

SUMMARY:
A. To evaluate the ocular hypotensive efficacy of the rho-kinase Inhibitor (AR-12286 0.5% and 0.7%) ophthalmic solutions in glaucoma patients with failed prior glaucoma filtering surgery and uncontrolled IOP who are facing further surgical intervention. Patients will be treated for 6 months in this initial trial.

B. To evaluate the efficacy of AR-12286 in enabling treated patients to delay or avoid the necessity of further surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years of either sex.
2. Patients with open-angle glaucoma with prior glaucoma filtering surgery.
3. IOP above the target range or visual field progression.
4. Have given written informed consent, prior to any investigational procedures.
5. Ability to attend for the 6-month duration of treatment.

Exclusion Criteria:

1. Closed angle glaucoma (primary or secondary).
2. Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
3. Ocular medication of any kind within 30 days of base-line visit, with the exception of ocular hypotensive medications and/or lubricating drops for dry eye (which may be used throughout the study).
4. Any abnormality preventing reliable applanation tonometry of the treated eye.
5. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
6. Participation in any investigational study within the past 30 days.
7. Inability to perform reliable visual field testing.
8. Unwilling to sign the consent form approved by the Institutional Review Board (IRB) of the New York Eye and Ear Infirmary.
9. Self-reported poor compliance to treatment.
10. Reluctance to return for scheduled follow-up visits.
11. Patients not able to understand the nature of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Effect of study drug to reduce IOP | 6 Months
  To evaluate the ocular hypotensive efficacy of Rho Kinase Inhibitor (AR-12286 0.5% and 0.7%) ophthalmic solutions in patients with uncontrolled Advanced Glaucoma with Prior Failed Trabeculectomy or Tube Shunt. The long lasting effect of the AR-12286 drug is hoped to increase aqueous outflow and clear the trabecular meshwork of material and reduce IOP.

SECONDARY OUTCOMES:
IOP Reduction | 6 Months
  To determine if AR-12286 can be used as directed therapy for Advanced Glaucoma with Prior Failed Trabeculectomy or Tube Shunt to avoid additional surgical intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Associates of New York, New York, New York, United States